CLINICAL TRIAL: NCT02640872
Title: A Hospital-based Prospective Cohort Study With Aged People to Elucidate Predictive Factors Including Muscle and Fat Mass for Chronic Diseases and Mortality
Brief Title: A Prospective Cohort Study of Aged People for Chronic Diseases
Acronym: HAPPY
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, MD, PhD, Seoul National University Bundang Hospital
Other Study IDs: SNUBH-HAPPY Cohort
Record Dates: First submitted 2015-12-19; First posted 2015-12-29 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Aging; Sarcopenia
Keywords: sarcopenia; sarcopenic obesity; osteoporosis; fracture; cardiovascular disease; mortality
MeSH Terms: conditions — Sarcopenia; Osteoporosis; Fractures, Bone; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — for measuring biomarkers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HAPPY Cohort: A elderly cohort for chronic diseases

SUMMARY:
This study is a hospital-based, prospective cohort study to elucidate the predictive factors including muscle and fat mass for chronic diseases and mortality in elderly persons aged 60 years and older.

DETAILED DESCRIPTION:
This study is a hospital-based, prospective cohort study to elucidate the predictive factors among anthropometric and biochemical parameters and body composition information for chronic diseases including diabetes mellitus, myocardial infarction, stroke, osteoporosis, fracture, and cognitive dysfunction, and mortality in elderly persons aged 60 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and older
* Capable of communication with the research team
* Provided written informed consent

Exclusion Criteria:

* Age < 60 years
* active malignancy
* uncompensated liver cirrhosis
* ESRD
* severe cognitive impairment which cannot communicate with the research term

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aged 60 years and older Capable of communication with the research team Provided written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Alll cause mortality | 9 years

SECONDARY OUTCOMES:
Cardiometabolic mortality | 9 years
Incidence of major adverse cardiac event including nonfatal myocardial infarction, nonfatal stroke, and unstable angina | 9 years
Incidence of frailty defined by the Korean Fraility Index | 9 years
Incidence of osteoporotic fracture | 9 years
Incidence of cognitive dysfunction measured by minimental status examination | 9 years
Development of sarcopenia defined by the Foundation for the National Institutes of Health (FNIH) criteria | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — SNUBH
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No